CLINICAL TRIAL: NCT05239390
Title: Phase IIA Open-Label, to Evaluate the Safety, Tolerability, and Efficacy Trend of SCI -110 in Patients With AD and Agitation
Brief Title: SCI-110 for Alzheimer Disease and Agitation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Israeli Medical Center for Alzheimer's (Other)
Responsible Party: Principal Investigator, dr. Alexander Kaplan, Principal Investigator, The Israeli Medical Center for Alzheimer's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAVE-Sci-001
Record Dates: First submitted 2021-07-25; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Dronabinol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCI -110 (Experimental): SCI -110 (Previously known as THX-110): a combination of THC (Doses: 2.5 mg - 12.5 mg per daily dose) and PEA (Dose: 800 mg per daily dose), administered together as separate pills, orally, twice daily (morning and evening - except for the initial titration dose, of 2.5 mg THC+800 mg PEA given once a day, in the morning.
  Interventions: Drug: SCI -110

INTERVENTIONS:
Drug: SCI -110 — Dronabinol - Manufactured by Pharmaceutics International, Inc., Hunt Valley, MD 21031, USA. Dronabinol Capsules (dronabinol solution in sesame oil in soft gelatin capsules) are 2.5 mg - cream, oblong, soft-gel capsules. In an NDC 49884-867-02 Bottle of 60 capsules packaged in a well-closed container and stored in a locked refrigerator, 2° to 8°C. Protect from freezing, in accordance with the Israeli legal requirements (Israel Narcotic Drugs Act). Storage conditions should be monitored on a daily basis.
  PEA - Manufactured by Pharmacies Inc. 767 Front st. Suite 202. Catasauqua, PA 18032 www.pharmacures.com. 1-888-334-3130. 400 mg PEA tablets, in a 60 mL barrier bottle, 30/400 mm, Bottle of 30 capsules packaged in a well-closed container and stored in RT (20° to 25°C). Storage conditions should be monitored on a daily basis.
  Other Names: Dronabinol and PEA

SUMMARY:
As of today, there is no FDA-approved treatment for agitation in AD. Hence, it is still considered an unmet need.

Sporadic observation in healthy or diagnosed individuals indicated that cannabis products, in particular, THC have calming and anti-anxiety effects. These observations are supported by basic science data as well as animal experiments.

SCI -110 is a combination of (1) dronabinol, the active ingredient in an FDA-approved synthetic analog of tetrahydrocannabinol, the psychoactive molecule in the cannabis plant, and (2) palmitoylethanolamide.

In the present study, the starting daily dose for all subjects is 2.5 mg dronabinol and 800 mg PEA and will be gradually increased (every 3 days an addition of 2.5 mg dronabinol per day, with no change in the PEA dose) to a maximum of 12.5 mg Dronebinol and 800 mg PEA per day. The study product will be given orally, twice daily, to add-on the medical treatment.

Study Duration per patient is up to 64 days: a. screening (3-21 days); b. treatment phase: (1) titration (15-23 days) of dronabinol from 2.5 to 12.5 mg or up to the maximal subject's tolerated dose (2) Stabilization phase (10 days) until end of treatment on the highest subject's daily tolerated dose. c. follow-up phase (7 days) - until the end-of-study.

During the study, the tolerability of the drug, its safety (vital signs, physical examinations, blood, and urine tests and side effects follow-up) as well as changes in subject's condition (using CMAI, MMSE, SIB-8 questionnaires), appetite and sleep quality (SDI) will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >60 to <85 years inclusive.
* Patients diagnosed according to the NINCDS criteria for AD (possible and probable).
* MMSE less than 24 at the time of screening.
* Patients who in the opinion of the investigators need medication to control agitation or whose current anti-agitation medication is ineffective or poorly tolerated
* Patients who have been taking stable dose concomitant medications for at least 1 week.
* Only individuals who have a legally appointed guardian who can sign Informed Consent Form (ICF)

Exclusion Criteria:

* Participant in other clinical trial during the last 30 days.
* Any disorder which in the investigator's opinion might jeopardize subject's safety or compliance with the protocol.
* Patients whose agitation can be attributed to a somatic disorder (Ex. urinary tract infection or urinary retention)
* Patient with uncontrolled congestive heart failure.
* Patients who get the following medications: opiates, Primidone, Phenobarbitol, carbamazepine, Rifampicin, Rifabutin, Troglitazone and Hypericum perforatum.
* Male patients who in the opinion of the investigator are at risk of urinary retention due to the anticholinergic proprieties of THC
* Subjects with known sensitivity to the active substance dronabinol or to any of the components of the drug (sesame oil, gelatin, glycerol, titanium dioxide
* Subjects that previously suffered from cannabinoids' related adverse effects.
* Subjects with a history of diagnosed Mental or Psychiatric diseases
* Patients who in the opinion of the investigator are at risk of falling beyond the risk associated with AD (example: postural hypotension, unstable blood pressure, with or without administration of anti-hypertensive medication, α1 blocker drugs used to treat benign prostatic hyperplasia
* Patients diagnosed with epilepsy

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-06-29 (Estimated); Study Completion 2023-06-29 (Estimated)

PRIMARY OUTCOMES:
drop-out's | up to 64 days
  Number of drop-out subjects' due to poor tolerability
Adverse Events | up to 64 days
  Number of study treatment (SCI -110) related Adverse Events (AEs) from Baseline (visit 2, day 1) to end of treatment.

SECONDARY OUTCOMES:
Change in the Cohen Mansfield Agitation Inventory (CMAI). | up to 64 days
  Change from Baseline to end of treatment in agitation measured by the Cohen Mansfield Agitation Inventory (CMAI).
rescue medication | up to 64 days
  Frequency of use of rescue medication to control agitation (Frequency of rescue medication use = number of drug administration(s) regardless of dose
Change in Mini Mental State Exam (MMSE) | up to 64 days
  Change from Baseline (visit 2, day 1) to end of treatment in Mini Mental State Exam (MMSE)
Change in Sleep Disorders Inventory | up to 64 days
  Change in quality of sleep from Baseline (visit 2, day 1) to end of treatment measured in Sleep Disorders Inventory
Change in The Edinburgh Feeding Evaluation in Dementia Scale | up to 64 days
  Change in appetite from Baseline (visit 2, day 1) to end of treatment measured in The Edinburgh Feeding Evaluation in Dementia Scale
Change in cognitive measures from Baseline (visit 2, day 1) to end of treatment measured in SIB-8 8-item Severe Impairment Battery | up to 64 days
  Change in SIB-8 8-item Severe Impairment Battery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kaplan, Principal Investigator — The Israeli Medical Center for Alzheimer's
Locations (1):
- The Israeli Medical Center for Alzheimer's, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No